CLINICAL TRIAL: NCT05297500
Title: Accuracy of Pulse Oximeters With Profound Hypoxia NIHO 14
Brief Title: Determination of SpO2 and PR Accuracy Specifications at Rest (71Ag_Vital-0031)
Status: Active, not recruiting | Type: Observational
Sponsor: Nihon Kohden (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 71Ag_Vital-0031
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2024-11

CONDITIONS: Hypoxia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult healthy subjects: Adult healthy subjects capable of undergoing controlled hypoxemia to the levels outlined in the desaturation profile in an at rest state
  Interventions: Device: Pulse oximeter

INTERVENTIONS:
Device: Pulse oximeter — OLV-4202 pulse oximeter (SW version: 01-12)

SUMMARY:
The aim of this study is to determine the accuracy of devices called pulse oximeters, which measure blood oxygen by shining light through fingers, ears or other skin, without requiring blood sampling. Study will be used with patients at rest

DETAILED DESCRIPTION:
This study is intended to evaluate performance of a new design pulse oximeter (test device) manufactured by Nihon Kohden Corporation sufficiently to support performance claims for an FDA 510K submission or ISO technical file. Specifically, SpO2 and pulse rate accuracy will be assessed for a Nihon Kohden OLV-4202 pulse oximeter with adult patients under a controlled setting of varying levels of inhaled oxygen concentration levels for patients at rest.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects who can give written informed consent
* Healthy subjects capable of undergoing controlled hypoxemia to the levels outlined in the desaturation profile
* Meeting the demographic requirements

Exclusion Criteria:

* Pregnant women
* Significant arrhythmia
* Blood pressure above 150 systolic or 90 diastolic
* Carboxyhemoglobin levels over 3%
* Subjects whom the investigator consider ineligible for the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers. At least 10 subjects will be recruited to complete the study. Of these 2 will be dark pigmented. If the number of samples is less than the required 200 or if less than 2 of dark pigment subjects successfully complete the study, subjects will be added to include 2 of dark pigmented subjects and at least 200 data points.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2026-10-29 (Estimated)

PRIMARY OUTCOMES:
Root-mean-square (Rms) of device SpO2 measurement with room air stabilization is within +-2% [%SpO2] of reference co-oximeter SaO2 measurement at varying desaturation levels (70% to 100%) | 30 minutes
  Each subject will have an arterial catheter inserted in the left or right wrist and the pulse oximeter study device placed on different fingers of the left or right hand, or the left or right earlobe or the forehead. Measurement position is randomized across subjects. For each subject, a series of desaturation runs are performed.
  Run 1 stabilized room air period -> stabilized plateaus at saturation level targets:
  room air, 92%, 87%, 82%, 77%, 72%
  Run 2 stabilized 100% O2 period -> stabilized plateaus at saturation level targets:
  100%, 93%, 88%, 83%, 78%, 73%
  SpO2 is observed breath by breath arterial saturation, which is in turn computed from end tidal PO2 and PCO2. FiO2 is reduced suddenly at first then adjusted to achieve a stable plateau value at the desired target. Each desaturation plateaus should not exceed 10 minutes. A blood draw is taken at stable FiO2 and +30 seconds. The gas mixture is then changed for the next value and repeated for each plateau value.
Root-mean-square (Rms) of device Pulse Rate measurement with room air stabilization is within +-3 [1/min] of reference ECG Pulse Rate measurement at heart rates (30 to 300 [1/min]) | 30 minutes
  Each subject will have an arterial catheter inserted in the left or right wrist and the pulse oximeter study device placed on different fingers of the left or right hand, or the left or right earlobe or the forehead. Measurement position is randomized across subjects. For each subject, a series of desaturation runs are performed.
  Run 1 stabilized room air period -> stabilized plateaus at saturation level targets:
  room air, 92%, 87%, 82%, 77%, 72%
  Run 2 stabilized 100% O2 period -> stabilized plateaus at saturation level targets:
  100%, 93%, 88%, 83%, 78%, 73%
  Pulse rate is recorded from the test device and from the reference ECG monitor. PR data measurements are gathered during the stable plateau value at the desired saturation target. Each desaturation plateaus should not exceed 10 minutes. The gas mixture is then changed for the next value and repeated for each plateau value.

SECONDARY OUTCOMES:
Root-mean-square (Rms) of device SpO2 measurement with room air stabilization is within +-2% [%SpO2] of reference co-oximeter SaO2 measurement at desaturation levels (80% to 100%) and within +-3% [%SpO2] at desaturation levels (70% to 80%) | 30 minutes
  Each subject will have an arterial catheter inserted in the left or right wrist and the pulse oximeter study device placed on different fingers of the left or right hand, or the left or right earlobe or the forehead. Measurement position is randomized across subjects. For each subject, a series of desaturation runs are performed.
  Run 1 stabilized room air period -> stabilized plateaus at saturation level targets:
  room air, 92%, 87%, 82%, 77%, 72%
  Run 2 stabilized 100% O2 period -> stabilized plateaus at saturation level targets:
  100%, 93%, 88%, 83%, 78%, 73%
  SpO2 is observed breath by breath arterial saturation, which is in turn computed from end tidal PO2 and PCO2. FiO2 is reduced suddenly at first then adjusted to achieve a stable plateau value at the desired target. Each desaturation plateaus should not exceed 10 minutes. A blood draw is taken at stable FiO2 and +30 seconds. The gas mixture is then changed for the next value and repeated for each plateau value.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Hypoxia Research Laboratory, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Data to be used by Sponsor only

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05297500/Prot_SAP_000.pdf